CLINICAL TRIAL: NCT07219420
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study With Open-Label Extension to Evaluate the Efficacy and Safety of Bimekizumab in Study Participants With Palmoplantar Pustulosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Study Participants With Palmoplantar Pustulosis
Acronym: BeSeen
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPP001; U1111-1322-7183 (Registry Identifier: WHO universal trial number (UTN))
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Palmoplantar Pustulosis
Keywords: Bimekizumab, PPP
MeSH Terms: conditions — Psoriasis; Aggressive Periodontitis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab (Experimental): Subjects randomized to this arm will receive the bimekizumab dosing regimen for the entire duration of the study.
  Interventions: Drug: Bimekizumab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo during the initial treatment period before transitioning to bimekizumab in the maintenance treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Study participants will receive bimekizumab at pre-specified time points.
  Other Names: BIMZELX, UCB4940
  Arms: Bimekizumab
Drug: Placebo — Study participants will receive matching placebo at pre-specified time points.
  Other Names: PLB
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of bimekizumab compared with placebo in participants with palmoplantar pustulosis (PPP).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age inclusive, at the time of signing the informed consent form (ICF)
* Have a palmoplantar pustulosis (PPP) diagnosis for at least 24 weeks prior to the Screening Visit
* Have PPPASI ≥12 at the Screening Visit and Baseline Visit
* Have PPP-IGA ≥3 at the Screening Visit and Baseline Visit
* Have pustules on the palms of the hands and/or soles of the feet at the Screening Visit and Baseline Visit, defined as pustule severity ≥2 and having more than 5 active pustules
* Participant must be a candidate for systemic therapy or phototherapy

Exclusion Criteria:

* Has PPP symptoms which improve significantly between the Screening Visit and Baseline Visit, defined as a reduction in the PPPASI score
* Has the following: palmoplantar PSO (plaque PSO on palms/soles), guttate PSO, erythrodermic PSO (EP), generalized pustular PSO (GPP), Acrodermatitis continua of Hallopeau (ACH), atopic dermatitis, dyshidrotic eczema or chronic hand eczema.
* Has drug-induced PSO (eg, first onset or current exacerbation due to beta blockers, calcium channel inhibitors, lithium, or tumor necrosis factor [TNF] inhibitor) or drug-induced pustular PSO (eg, acute generalized exanthematous pustulosis, acute localized exanthematous pustulosis)
* Has cutaneous lesions that may interfere with the evaluation of the affected area and/or evaluation of the severity of PPP
* Is taking or has taken prohibited or restricted medications without meeting the mandatory discontinuation or stability period relative to the Baseline Visit
* Is taking or has ever taken an interleukin (IL)-17A/IL-17F inhibitor, including bimekizumab, or has participated in a bimekizumab investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-12-27 (Estimated); Study Completion 2029-10-29 (Estimated)

PRIMARY OUTCOMES:
Palmoplantar pustulosis-Investigator Global Assessment 0/1 (PPP-IGA 0/1) response at Week 16 | At Week 16
  PPP-IGA is an overall assessment by a physician regarding condition of skin lesions on the palms and the soles in PPP. The Investigator will assess the overall severity of PPP using the following 5-point scale: 0 = Clear; 1 = Almost clear; 2 = Mild ; 3 = Moderate; 4 = Severe.

SECONDARY OUTCOMES:
Palmoplantar Pustulosis Area Severity Index 50 (PPPASI50) response at Week 16 | At Week 16
  The PPPASI50 response is based on at least 50% improvement from baseline in the PPPASI total score which assesses the severity of PPP skin lesions.
  The PPPASI evaluates 4 areas: right palm, left palm, right sole, and left sole which account for 20%, 20%, 30%, and 30%, respectively, of the total surface area of the palms or soles. Each palm and sole is evaluated for 3 characteristics:
  erythema, pustule, and desquamation. Each characteristic is rated on a 5-point severity scale, from 0 (none) to 4 (very severe). The percentage of area affected by PPP skin lesions is also evaluated for each palm and sole.
  The PPPASI total score ranges from 0 to 72, with a higher score indicating higher disease severity.
PPPASI75 response at Week 16 | At Week 16
  The PPPASI75 response is based on at least 75% improvement from baseline in the PPPASI score.
PPPASI90 response at Week 16 | At Week 16
  The PPPASI90 response is based on at least 90% improvement from baseline in the PPPASI score.
PPPASI50 response at Week 8 | At Week 8
  The PPPASI50 response is based on at least 50% improvement from baseline in the PPPASI score.
PPP-IGA 0/1 response at Week 8 | At Week 8
  PPP-IGA is an overall assessment by a physician regarding condition of skin lesions on the palms and the soles in PPP.
Change from Baseline in Dermatology Life Quality Index (DLQI) total score at Week 16 | From Baseline to Week 16
  The DLQI is a skin disease-specific questionnaire aimed at the evaluation of how symptoms and treatment affect participants' health-related quality of life (HRQOL). This questionnaire asks participants 10 questions about symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. For each question, participants are asked to evaluate on a 4-point scale (from 0=Not at all to 3=Very much) to which extend their skin disease has affected their life over the last week. The DLQI total score ranges from 0 to 30 with higher scores indicating lower HRQOL.
Change from Baseline in Numerical Rating Scale (NRS) - PPP Pain score in the palmoplantar areas at Week 16 | From Baseline to Week 16
  The study participant will score the worst level of PPP skin pain over the past 24 hours on a 11-point NRS from "0=no skin pain" to "10=very severe skin pain.
Incidence of treatment-emergent adverse events (TEAEs) from Baseline to the end of the Safety Follow-up (SFU) Period | From Baseline (Day 1) until Safety Follow-Up (up to Week 112)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 12 weeks.
Incidence of serious TEAEs from Baseline to the end of the SFU Period | From Baseline (Day 1) until Safety Follow-Up (up to Week 112)
  An SAE is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 12 weeks.
Incidence of TEAEs leading to permanent discontinuation of study treatment from Baseline to the end of the SFU Period | From Baseline (Day 1) until Safety Follow-Up (up to Week 112)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Treatment-emergent AEs are defined as those AEs that have a start date on or following the first dose of IMP through the final dose of IMP + 12 weeks. This measure considers any TEAE leading to permanent discontinuation of IMP regardless of reason.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 22733 (UCB)
Locations (14):
- Canada (2):
  - Ppp001 50233, Barrie
  - Ppp001 50740, Québec
- China (6):
  - Ppp001 20137, Chengdu
  - Ppp001 20350, Chongqing
  - Ppp001 20313, Guangzhou
  - Ppp001 20022, Hangzhou
  - Ppp001 20345, Shanghai
  - Ppp001 20184, Shenzhen
- Ppp001 40875, Ahaus, Germany
- Hungary (2):
  - Ppp001 40895, Debrecen
  - Ppp001 40894, Orosháza
- Poland (3):
  - Ppp001 40625, Lodz
  - Ppp001 40604, Warsaw
  - Ppp001 40862, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org